CLINICAL TRIAL: NCT00077558
Title: A Phase I Trial Of Sequential Administration Of Triapine (3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone) Followed By Fludarabine In Adults With Relapsed And Refractory Leukemias And Myelodysplasias
Brief Title: 3-AP Followed By Fludarabine In Treating Patients With Relapsed or Refractory Acute or Chronic Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000352322, J0357; U01CA070095 (NIH); P30CA006973 (NIH); JHOC-J0357; NCI-6255
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory chronic lymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; prolymphocytic leukemia; refractory anemia with excess blasts; chronic myelomonocytic leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute promyelocytic leukemia (M3); adult acute eosinophilic leukemia; adult acute basophilic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — fludarabine phosphate; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: fludarabine phosphate
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. 3-AP may help fludarabine kill more cancer cells by making them more sensitive to the drug.

PURPOSE: This phase I trial is studying the side effects and best dose of fludarabine when given together with 3-AP in treating patients with relapsed or refractory acute leukemia, chronic leukemia, or high-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and tolerability of 3-AP (Triapine^® ) followed by fludarabine in patients with relapsed or refractory acute or chronic leukemia or high-risk myelodysplastic syndromes.
* Determine the toxic effects of this regimen in these patients.
* Determine the maximum tolerated dose of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of fludarabine. Patients are stratified according to disease (acute leukemias and myelodysplastic syndromes [MDS] vs chronic lymphocytic leukemia and prolymphocytic leukemia). Patients are assigned to 1 of 2 treatment groups.

* Group 1 (chronic lymphocytic leukemia or prolymphocytic leukemia): Patients receive 3-AP (Triapine^®) IV over 4 hours and fludarabine IV over 30 minutes on days 1-5.

Cohorts of 3-6 patients receive escalating doses of fludarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at that dose level.

* Group 2 (acute leukemias or MDS): Patients receive 3-AP IV continuously over 24 hours on day 1. Beginning within 4 hours after completion of 3-AP, patients receive fludarabine IV over 30 minutes on days 2-6.

In both groups, treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 3-34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * High-risk myelodysplastic syndromes (MDS), including refractory anemia with excess blasts and chronic myelomonocytic leukemia

    * International Prognostic Scoring System (IPSS) score at least 1.5 based on the following:

      * More than 10% marrow blasts
      * Cytopenias in at least 2 lineages
      * Adverse cytogenetics
  * Acute myeloid leukemia (AML)

    * All subtypes, including MDS/AML and treatment-related (secondary) AML
  * Acute lymphoblastic leukemia
  * Acute progranulocytic leukemia

    * Ineligible for arsenic therapy
  * Chronic myelogenous leukemia

    * Accelerated phase or blastic crisis
  * Chronic lymphocytic leukemia
  * Prolymphocytic leukemia
* Received or ineligible for established curative regimens, including stem cell transplantation
* Acute and chronic leukemias must be relapsed and/or refractory with progressive disease since last therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* No history of hemolytic anemia grade 2 or greater
* No known glucose-6-phosphate dehydrogenase (G6PD) deficiency

  * G6PD screening required for high-risk groups (i.e., patients of African, Asian, or Mediterranean origin/ancestry)

Hepatic

* SGOT and SGPT no greater than 2.5 times normal
* Bilirubin no greater than 2 mg/dL
* No chronic hepatitis

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No active heart disease
* No myocardial infarction within the past 3 months
* No severe coronary artery disease
* No arrhythmias (other than atrial flutter or fibrillation) requiring medication
* No uncontrolled congestive heart failure

Pulmonary

* No dyspnea at rest or with minimal exertion
* No severe pulmonary disease requiring supplemental oxygen

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy grade 2 or greater
* No active uncontrolled infection

  * Infections under active treatment and controlled by antibiotics are allowed
* No other life-threatening illness
* No psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 1 week since prior hematopoietic growth factor (e.g., epoetin alfa, filgrastim [G-CSF], sargramostim [GM-CSF], interleukin-3, and interleukin-11)
* No concurrent immunotherapy

Chemotherapy

* Recovered from prior chemotherapy (no greater than grade 1 chronic toxic effects)
* At least 72 hours since prior hydroxyurea
* At least 3 weeks since prior myelosuppressive cytotoxic agents (6 weeks for mitomycin or nitrosoureas)
* No more than 12 prior courses of fludarabine
* No more than 3 prior cytotoxic chemotherapy regimens
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 1 week since prior non-myelosuppressive treatment
* No more than 4 prior induction regimens
* No other concurrent therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (4):
- United States (4):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Karp JE, Giles FJ, Gojo I, Morris L, Greer J, Johnson B, Thein M, Sznol M, Low J. A phase I study of the novel ribonucleotide reductase inhibitor 3-aminopyridine-2-carboxaldehyde thiosemicarbazone (3-AP, Triapine) in combination with the nucleoside analog fludarabine for patients with refractory acute leukemias and aggressive myeloproliferative disorders. Leuk Res. 2008 Jan;32(1):71-7. doi: 10.1016/j.leukres.2007.05.003. Epub 2007 Jul 20. PMID 17640728